CLINICAL TRIAL: NCT04299295
Title: A Study to Evaluate the Performance and Safety of YVOIRE Y-Solution 360 Versus Comparator for Temporary Enhancement and Pouting of the Lips for Lip Augmentation and Correction of Perioral Area.
Brief Title: To Evaluate the Performance and Safety of YVOIRE Y Solution 360 Versus Comparator for Lips and Perioral Area.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to company's internal decision.
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LG-HACL023
Record Dates: First submitted 2020-03-02; First posted 2020-03-06 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2020-06

CONDITIONS: Lip Augmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YVOIRE Y-Solution 360 (Experimental): Hyaluronic acid dermal filler
  Interventions: Device: YVOIRE Y-Solution 360
- Juvéderm VOLBELLA (Active Comparator): Hyaluronic acid dermal filler
  Interventions: Device: Juvéderm VOLBELLA

INTERVENTIONS:
Device: YVOIRE Y-Solution 360 — Hyaluronic acid dermal filler
  Arms: YVOIRE Y-Solution 360
Device: Juvéderm VOLBELLA — Hyaluronic acid dermal filler
  Arms: Juvéderm VOLBELLA

SUMMARY:
A Study to Evaluate the Performance and Safety of YVOIRE Y-Solution 360 on Lips and Perioral Area.

DETAILED DESCRIPTION:
This is a Randomized, Multicenter, Evaluator-Blinded, Active-Controlled, Parallel-Group Study to Evaluate the Performance and Safety of YVOIRE Y-Solution 360 Versus Comparator for Temporary Enhancement and Pouting of the Lips for Lip Augmentation and Correction of Perioral Area

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or above age.
* 1 or 2 of the 5-point (0-4) LFRS (Lip Fullness Rating Scale).
* Agree to use proper contraception as guided in the protocol.
* Signed for Informed Consent.

Exclusion Criteria:

* have lip tattoos, piercings, facial hair, or scars that would interfere with visualization of the lips and perioral area
* who have dentures or any device covering all or part of the upper palate, and/or severe malocclusion or dentofacial or maxillofacial deformities
* have undergone oral surgery within 6 weeks
* have received permanent facial implants in the face or neck, or are planning to be implanted with any of these products
* have undergone semi-permanent filler in lower face within 24 months
* have undergone temporary dermal filler treatment in the lower face within 12 months
* Have undergone facial tissue augmentation or facial treatment with fat or botulinum injections in the lower face within 6 months
* Have undergone mesotherapy, face lift, laser, photo modulation, intense pulsed light, radio frequency, dermabrasion, moderate or greater depth chemical peel, or other ablative procedures in face or neck within 6 months
* have used lip plumping products within 10 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Mean change on the overall Lip Fullness Rating Scale (LFRS) from baseline to Week12. | 12 weeks from baseline
  To evaluate the performance of YVOIRE Y-Solution 360 on overall Lip 12 weeks after treatment, the mean change from baseline to 12 weeks will be measured using 5-point Lip Fullness Rating Scale (LFRS). LFRS Grades are 0 (None/Minimal), 1 (Mild), 2 (Moderate), 3 (Pronounced), and 4 (Very Pronounced).
Responder rate calculated using Lip Fullness Rating Scale (LFRS) for overall lip at Week12. | 12 weeks from baseline
  To evaluate the performance of YVOIRE Y-Solution 360 on overall Lip 12 weeks after treatment, the responder rate defined as ≥ 1-point improvement on the 5-point Lip Fullness Rating Scale (LFRS) from baseline to 12 weeks will be calculated.

SECONDARY OUTCOMES:
Mean change on Lip Fullness Rating Scale (LFRS) from baseline to Week2, 4, 12 and 24. | 2, 4, 12, 24 weeks from baseline
  To evaluate the performance of YVOIRE Y-Solution 360 at 2, 4, 12, and 24 weeks after treatment, the mean change from baseline to at 2, 4, 12, and 24 weeks will be measured using 5-point Lip Fullness Rating Scale (LFRS).
Responder rate on Lip Fullness Rating Scale (LFRS) from baseline to Week2, 4, 12 and 24. | 2, 4, 12, 24 weeks from baseline
  To evaluate the performance of YVOIRE Y-Solution 360 at 2, 4, 12, and 24 weeks after treatment, the responder rate (defined as at a least 1-point improvement) from baseline to at 2, 4, 12, and 24 weeks will be measured using 5-point Lip Fullness Rating Scale (LFRS).
Mean change on Vertical Perioral Lip lines Rating Scale - At rest(VPLRS) from baseline to Week2, 4, 12 and 24. | 2, 4, 12, 24 weeks from baseline
  To evaluate the performance of YVOIRE Y-Solution 360 on perioral area at 2, 4, 12, and 24 weeks after treatment, the mean change from baseline to at 2, 4, 12, and 24 weeks will be measured using 5-point Vertical Perioral Lip lines Rating Scale - At rest (VPLRS).
Responder rate on Vertical Perioral Lip lines Rating Scale - At rest(VPLRS) from baseline to Week2, 4, 12 and 24. | 2, 4, 12, 24 weeks from baseline
  To evaluate the performance of YVOIRE Y-Solution 360 on perioral area at 2, 4, 12, and 24 weeks after treatment, the responder rate (as at a least 1-point improvement) from baseline to at 2, 4, 12, and 24 weeks will be measured using 5-point Vertical Perioral Lip lines Rating Scale - At rest (VPLRS).
Global Aesthetic Improvement Scale (GAIS) evaluation by subject and investigator. | 2, 4, 12, 24 weeks from baseline
  To measure the satisfaction of YVOIRE Y-Solution 360 the GAIS evaluation will be performed by subject and investigator. GAIS Grade are -2 (Much Worse), -1 (Worse), 0 (No change), 1 (Improved), and 2 (Much improved).

CONTACTS AND LOCATIONS:
Overall Officials: Tanja C. Fischer, Principal Investigator — Haut-und Lasercentrum Potsdam
Locations (1):
- Haut-und Lasercentrum Potsdam, Potsdam, Germany

IPD SHARING:
Plan to Share IPD: No